CLINICAL TRIAL: NCT00349193
Title: A Multinational, Multicenter Randomized Double-Blind, Parallel-Group, Placebo-Controlled Study, to Evaluate the Efficacy, Tolerability and Safety of Two Doses of, Oral Laquinimod in Relapsing Remitting (R-R) Multiple Sclerosis (MS) Subjects
Brief Title: A Study to Evaluate the Effectiveness, Tolerability and Safety of Laquinimod
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Ekkehard Baader, MD, Teva Pharmaceutical Europe B.V.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAQ/5062; 2004-003943-28 (EudraCT Number)
Record Dates: First submitted 2006-06-26; First posted 2006-07-06 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2011-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laquinimod 0.3 mg (Active Comparator): Laquinimod 0.3 mg
  Interventions: Drug: laquinimod 0.3
- Laquinimod 0.6 mg (Active Comparator): Laquinimod 0.6 mg
  Interventions: Drug: laquinimod 0.6
- Placebo (Placebo Comparator): Blinded Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: laquinimod 0.3 — laquinimod 0.3mg
  Arms: Laquinimod 0.3 mg
Drug: laquinimod 0.6 — laquinimod 0.6mg
  Arms: Laquinimod 0.6 mg
Other: Placebo — Blinded Placebo
  Arms: Placebo

SUMMARY:
Teva is developing laquinimod tablets as a new oral treatment for MS. Laquinimod has immunomodulating properties. In a previous clinical study laquinimod showed evidence of biological activity by reducing the number of acute brain lesions.

The duration of the current study is 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent
2. Confirmed MS diagnosis as defined by the McDonald criteria
3. R-R MS disease course.
4. At least one gadolinium-enhanced lesion on screening MRI
5. Women of child-bearing potential must practice a reliable method of birth control.
6. Must understand the requirements of the study and agree to comply with the study protocol.

Exclusion Criteria:

1. Subjects who suffer from any form of progressive MS.
2. Any condition which the investigator feels may interfere with participation in the study.
3. Subjects with a clinically significant or unstable medical or surgical condition that would preclude safe and complete study participation,
4. Subjects who received any investigational medication, immunosuppressives or cytotoxic agents within 6 months prior to screening
5. Previous treatment with immunomodulators within two months prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Reduction of brain lesions in the last 4 months of the study | 36 weeks

SECONDARY OUTCOMES:
Relapse rate | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Giancarlo Comi, Study Chair — Teva Pharmaceutical Industries, Ltd.

REFERENCES:
- [Derived] Comi G, Pulizzi A, Rovaris M, Abramsky O, Arbizu T, Boiko A, Gold R, Havrdova E, Komoly S, Selmaj K, Sharrack B, Filippi M; LAQ/5062 Study Group. Effect of laquinimod on MRI-monitored disease activity in patients with relapsing-remitting multiple sclerosis: a multicentre, randomised, double-blind, placebo-controlled phase IIb study. Lancet. 2008 Jun 21;371(9630):2085-92. doi: 10.1016/S0140-6736(08)60918-6. PMID 18572078